CLINICAL TRIAL: NCT04870255
Title: Modulating Probabilities: Prediction, Assessment, and Treatment of Acute Mood Depressive Episode in Borderline Personality Disorder With rTMS
Brief Title: Treatment of Acute Mood Depressive Episode in Borderline Personality Disorder With rTMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Spiegel, Professor, Psych/Major Laboratories and Clinical & Translational Neuroscience, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 58950
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Depressive Disorder, Major; Borderline Personality Disorder
Keywords: Depression; Neuromodulation; Transcranial Magnetic Stimulation; Borderline Personality Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Borderline Personality Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive: active L-DLPFC stimulation, active DMPFC stimulation, or sham stimulation. Group size ratio will be 1:1:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Left Dorsolateral Prefrontal Cortex (L-DLPFC) (Active Comparator): The accelerated theta burst stimulation protocol will be applied to the left dorsolateral prefrontal cortex (L-DLPFC)
  Interventions: Device: Left Dorsolateral Prefrontal Cortex (L-DLPFC)
- Dorsomedial Prefrontal Cortex (DMPFC) (Active Comparator): The accelerated theta burst stimulation protocol will be applied to the dorsomedial prefrontal cortex (DMPFC)
  Interventions: Device: Dorsomedial Prefrontal Cortex (DMPFC)
- Sham stimulation (Sham Comparator): Sham (non-active) stimulation will be applied to the left dorsolateral prefrontal cortex (DLPFC) region
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Left Dorsolateral Prefrontal Cortex (L-DLPFC) — Participants who are randomly assigned to this group will receive active iTBS (intermittent theta burst stimulation) to the left DLPFC. Stimulation intensity will be standardized at 90% of resting motor threshold (adjusted for cortical depth).
  Stimulation will be delivered using the Magventure Magpro X100 TMS system.
  Arms: Left Dorsolateral Prefrontal Cortex (L-DLPFC)
Device: Dorsomedial Prefrontal Cortex (DMPFC) — Participants who are randomly assigned to this group will receive active iTBS (intermittent theta burst stimulation) to the DMPFC. Stimulation intensity will be standardized at 100% of resting motor threshold (adjusted for cortical depth).
  Stimulation will be delivered using the Magventure Magpro X100 TMS system.
  Arms: Dorsomedial Prefrontal Cortex (DMPFC)
Device: Sham Stimulation — Participants who are randomly assigned to this group will receive sham stimulation to the left DLPFC.
  Sham stimulation will be delivered using the Magventure Magpro X100 TMS system.
  Arms: Sham stimulation

SUMMARY:
This study evaluates the antidepressant effects of an accelerated schedule of theta-burst stimulation, termed accelerated intermittent theta-burst stimulation (aiTBS), in individuals with borderline personality disorder (BPD) or trait and comorbid mood depressive disorder (MDD) or bipolar II disorder in a current mood depressive episode (MDE).

DETAILED DESCRIPTION:
This project aims to measure and modulate a mood depressive episode (MDE) in individuals with borderline personality disorder (BPD) trait and comorbid mood depressive disorder (MDD) or bipolar II disorder in a current mood depressive episode (MDE). This study will test the antidepressant effect of aiTBS stimulation over the left dorsolateral prefrontal cortex (L-DLPFC), and aiTBS stimulation over the dorsomedial prefrontal cortex (DMPFC) compared with sham.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, between the ages of 18 and 80 at the time of screening.
* Able to read, understand, and provide written, dated informed consent prior to screening. Proficiency in English sufficient to complete questionnaires / follow instructions during fMRI assessments and aiTBS interventions. Stated willingness to comply with all study procedures, including availability for the duration of the study, and to communicate with study personnel about adverse events and other clinically important information.
* Diagnosed with Major Depressive Disorder (MDD) or Bipolar II, or unspecified depressive disorder AND Borderline Personality Disorder or trait, with a current Mood Depressive Episode (MDE), according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5).
* MADRS score of ≥20 at screening (Visit 1).
* TMS naive.
* Access to ongoing psychiatric care before and after completion of the study.
* Access to clinical rTMS after study completion.
* In good general health, as evidenced by medical history.
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.
* Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration.

Exclusion Criteria:

* Pregnancy
* The presence or diagnosis of prominent anxiety disorder, personality disorder, or dysthymia
* Current severe insomnia (must sleep a minimum of 5 hours each night before stimulation)
* Current mania or psychosis
* Bipolar I Disorder and primary psychotic disorders.
* Autism Spectrum disorder or Intellectual Disability
* A diagnosis of obsessive-compulsive disorder (OCD)
* Current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal.
* Urine screening test positive for illicit substances.
* Any history of ECT (greater than 8 sessions) without meeting responder criteria
* Recent (during the current depressive episode) or concurrent use of a rapid acting antidepressant agent (i.e., ketamine or a course of ECT).
* History of significant neurologic disease, including dementia, Parkinson's or Huntington's disease, brain tumor, unexpected seizure/epilepsy disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma.
* Untreated or insufficiently treated endocrine disorder.
* Contraindications to receiving rTMS (e.g., metal in head, history of seizure, known brain lesion)
* Contraindications to MRI (ferromagnetic metal in their body).
* Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.
* Depth-adjusted aiTBS treatment dose > 65% maximum stimulator output (MSO)
* Treatment with another investigational drug or other intervention within the study period.
* Any other condition deemed by the PI to interfere with the study or increase risk to the participant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in the clinician rated Montgomery-Asberg Depression Rating Scale (MADRS-C) in active L-DLPFC vs. sham aiTBS. | At baseline (pre-intervention), during the intervention and immediately after the intervention.
  A ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.The MADRS-C has an overall score range from 0-60, with higher scores corresponding to higher levels of depression.

SECONDARY OUTCOMES:
Change in the clinician rated Montgomery-Asberg Depression Rating Scale (MADRS-C) in active DMPFC vs. sham aiTBS. | At baseline (pre-intervention), during the intervention and immediately after the intervention.
  A ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.The MADRS-C has an overall score range from 0-60, with higher scores corresponding to higher levels of depression.
Feasibility of aiTBS in individuals with BPD and comorbid MDD or BAD II in a current MDE as defined by retention rates | At baseline (pre-intervention), during the intervention and immediately after the intervention.
  Retention rates will be determined as research follow-up rate ≥80%
Feasibility of aiTBS in individuals with BPD and comorbid MDD or BAD II in a current MDE as defined by recruitment rate | At baseline (pre-intervention), during the intervention and immediately after the intervention.
  Recruitment rate will be determined by actual recruitment/recruitment milestones
Safety of aiTBS in individuals with BPD and comorbid MDD or BAD II in a current MDE as defined by rate of suicidal behaviors | At baseline (pre-intervention), during the intervention and immediately after the intervention.
  Rate of suicidal behaviors will be determined by number of participants that committed a SB/total number of participants

CONTACTS AND LOCATIONS:
Overall Officials: Nolan Williams, MD, Study Director — Stanford University; David Spiegel, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Background] Abdallah CG, Averill LA, Collins KA, Geha P, Schwartz J, Averill C, DeWilde KE, Wong E, Anticevic A, Tang CY, Iosifescu DV, Charney DS, Murrough JW. Ketamine Treatment and Global Brain Connectivity in Major Depression. Neuropsychopharmacology. 2017 May;42(6):1210-1219. doi: 10.1038/npp.2016.186. Epub 2016 Sep 8. PMID 27604566
- [Background] Liston C, Chen AC, Zebley BD, Drysdale AT, Gordon R, Leuchter B, Voss HU, Casey BJ, Etkin A, Dubin MJ. Default mode network mechanisms of transcranial magnetic stimulation in depression. Biol Psychiatry. 2014 Oct 1;76(7):517-26. doi: 10.1016/j.biopsych.2014.01.023. Epub 2014 Feb 5. PMID 24629537
- [Background] Green KL, Brown GK, Jager-Hyman S, Cha J, Steer RA, Beck AT. The Predictive Validity of the Beck Depression Inventory Suicide Item. J Clin Psychiatry. 2015 Dec;76(12):1683-6. doi: 10.4088/JCP.14m09391. PMID 26717528
- [Background] Ballard ED, Reed JL, Szczepanik J, Evans JW, Yarrington JS, Dickstein DP, Nock MK, Nugent AC, Zarate CA Jr. Functional Imaging of the Implicit Association of the Self With Life and Death. Suicide Life Threat Behav. 2019 Dec;49(6):1600-1608. doi: 10.1111/sltb.12543. Epub 2019 Feb 13. PMID 30761601
- [Background] Tello N, Harika-Germaneau G, Serra W, Jaafari N, Chatard A. Forecasting a Fatal Decision: Direct Replication of the Predictive Validity of the Suicide-Implicit Association Test. Psychol Sci. 2020 Jan;31(1):65-74. doi: 10.1177/0956797619893062. Epub 2019 Dec 11. PMID 31825760
- [Background] Light SN, Bieliauskas LA, Taylor SF. Measuring change in anhedonia using the "Happy Faces" task pre- to post-repetitive transcranial magnetic stimulation (rTMS) treatment to left dorsolateral prefrontal cortex in Major Depressive Disorder (MDD): relation to empathic happiness. Transl Psychiatry. 2019 Sep 3;9(1):217. doi: 10.1038/s41398-019-0549-8. PMID 31481688
- [Background] Baeken C, Duprat R, Wu GR, De Raedt R, van Heeringen K. Subgenual Anterior Cingulate-Medial Orbitofrontal Functional Connectivity in Medication-Resistant Major Depression: A Neurobiological Marker for Accelerated Intermittent Theta Burst Stimulation Treatment? Biol Psychiatry Cogn Neurosci Neuroimaging. 2017 Oct;2(7):556-565. doi: 10.1016/j.bpsc.2017.01.001. Epub 2017 Jan 20. PMID 29560909
- [Background] Downar J, Geraci J, Salomons TV, Dunlop K, Wheeler S, McAndrews MP, Bakker N, Blumberger DM, Daskalakis ZJ, Kennedy SH, Flint AJ, Giacobbe P. Anhedonia and reward-circuit connectivity distinguish nonresponders from responders to dorsomedial prefrontal repetitive transcranial magnetic stimulation in major depression. Biol Psychiatry. 2014 Aug 1;76(3):176-85. doi: 10.1016/j.biopsych.2013.10.026. Epub 2013 Nov 28. PMID 24388670
- [Background] Duprat R, De Raedt R, Wu GR, Baeken C. Intermittent Theta Burst Stimulation Increases Reward Responsiveness in Individuals with Higher Hedonic Capacity. Front Hum Neurosci. 2016 Jun 16;10:294. doi: 10.3389/fnhum.2016.00294. eCollection 2016. PMID 27378888
- [Background] Schmaal L, van Harmelen AL, Chatzi V, Lippard ETC, Toenders YJ, Averill LA, Mazure CM, Blumberg HP. Imaging suicidal thoughts and behaviors: a comprehensive review of 2 decades of neuroimaging studies. Mol Psychiatry. 2020 Feb;25(2):408-427. doi: 10.1038/s41380-019-0587-x. Epub 2019 Dec 2. PMID 31787757
- [Background] Gartner M, Aust S, Bajbouj M, Fan Y, Wingenfeld K, Otte C, Heuser-Collier I, Boker H, Hattenschwiler J, Seifritz E, Grimm S, Scheidegger M. Functional connectivity between prefrontal cortex and subgenual cingulate predicts antidepressant effects of ketamine. Eur Neuropsychopharmacol. 2019 Apr;29(4):501-508. doi: 10.1016/j.euroneuro.2019.02.008. Epub 2019 Feb 26. PMID 30819549